CLINICAL TRIAL: NCT05969093
Title: Refining the Interpretation of the Tinel's Sign for Carpal Tunnel Syndrome: An Electromyographic and Nerve Conduction Velocity Study
Brief Title: Refining the Interpretation of the Tinel's Sign for Carpal Tunnel Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Other Study IDs: 012/TINEL2023
Record Dates: First submitted 2023-07-22; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy individuals: Participants will undergo the Tinel's Sign at different wrist positions while EMG activity and NCV are recorded.
  Interventions: Diagnostic Test: Tinel's Sign performed at different wrist positions

INTERVENTIONS:
Diagnostic Test: Tinel's Sign performed at different wrist positions — Participants will undergo the Tinel's Sign at different wrist positions while EMG activity and NCV are recorded to investigate the effect of wrist position on median nerve activity.

SUMMARY:
This is an observational study to investigate the electromyographic (EMG) activity and nerve conduction velocity (NCV) of healthy individuals during the Tinel's Sign performed at different wrist positions. The study aims to identify the wrist position that best isolates median nerve activity during the Tinel's Sign.

DETAILED DESCRIPTION:
The study will be conducted in a controlled laboratory setting, equipped with an electromyography (EMG) machine and a nerve conduction velocity (NCV) measurement device. We will recruit 30 healthy adults, aged 18-45 years, with no history of hand or wrist pain, neurological or muscular disorders. Participants will be excluded if they have any contraindications to EMG or NCV measurement. The independent variable will be the wrist position during the Tinel's Sign, and the dependent variables will be the EMG activity of the thenar and hypothenar muscles and the NCV of the median and ulnar nerves. EMG activity will be measured using surface electrodes placed on the thenar and hypothenar muscles. NCV will be measured using a standard NCV measurement device. To minimize bias, the same trained examiner will perform all tests and measurements, and the examiner will be blinded to the EMG and NCV data during the tests. Differences in EMG activity and NCV across different wrist positions will be analyzed using repeated measures ANOVA. Post-hoc pairwise comparisons will be performed using Bonferroni correction. The study protocol will be submitted to the local ethics committee for approval, and all participants will provide informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals aged 18-45 years
* No history of hand or wrist pain, neurological or muscular disorders

Exclusion Criteria:

* Any contraindications to EMG or NCV measurement

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy individuals aged 18-60 years
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-07-29 (Estimated); Primary Completion 2023-12-23 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
EMG activity of the thenar muscles during the Tinel's Sign performed at different wrist positions. | Baseline
  The amplitude of EMG activity of the thenar muscles will be measured during the Tinel's Sign performed at different wrist positions. The amplitude will be quantified in microvolts (µV).
EMG activity of the hypothenar muscles during the Tinel's Sign performed at different wrist positions. | Baseline
  The amplitude of EMG activity of the hypothenar muscles will be measured during the Tinel's Sign performed at different wrist positions. The amplitude will be quantified in microvolts (µV).
Nerve conduction velocity of the median nerve during the Tinel's Sign performed at different wrist positions. | Baseline
  The NCV of the median nerve will be measured during the Tinel's Sign performed at different wrist positions. The NCV will be quantified in meters per second (m/s).
Nerve conduction velocity of the ulnar nerve during the Tinel's Sign performed at different wrist positions. | Baseline
  The NCV of the ulnar nerve will be measured during the Tinel's Sign performed at different wrist positions. The NCV will be quantified in meters per second (m/s).

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Chair — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No